CLINICAL TRIAL: NCT02704676
Title: CA-125 and Severity of Pre-Eclampsia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Bahaa Eldin Ahmed, Clinical professor, Ain Shams Maternity Hospital
Other Study IDs: CA125
Record Dates: First submitted 2016-03-03; First posted 2016-03-10 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-03

CONDITIONS: Pre-Eclampsia
Keywords: CA-125; Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- control patients: normal pregnant women, 3rd trimester
  Interventions: Other: marker(CA-125)
- mild pre-eclampsia: patients with albuminuria +1 and blood pressure >140/90 and <160/110
  Interventions: Other: marker(CA-125)
- sever pre-eclampsia: patients diagnosed as sever pre-eclampsia according to criteria done by ACOG
  Interventions: Other: marker(CA-125)

INTERVENTIONS:
Other: marker(CA-125) — measuring CA-125 in pregnant women (normal,mild and sever pre-eclampsia)

SUMMARY:
The Aim of this study is to determine the relationship between serum concentrations of cancer antigen-125 (CA-125) and pre-eclampsia severity.

DETAILED DESCRIPTION:
Although the source of CA-125 during pregnancy is the fetal chorion, amniotic fluid, and maternal decidua, the perinatal dynamics of maternal serum CA-125 requires clarification. Clinical studies of CA-125 levels and its function in hypertensive pregnant patients are limited and offered contradictory results (Cebesoy et al., 2009).

And so we investigate CA-125 in normal pregnancy and in pre-eclampsia, comparing mild and sever pre-eclampsia to determine relationship of CA-125 and severity of the disease.

Patients will be divided in three groups:

* Control: 40 normal healthy pregnant women attending the ER in labor.
* Mild pre-eclampsia: 40 patients fulfilling the following criteria.

  * Blood pressure: systolic blood pressure >140 and <160 , Diastolic blood pressure >90 and <110
  * Proteinuria: 300 mg (+) assessed by urine urignost 3A® (urine strips from DIALAB).
  * No symptoms of severity as headache.
  * Normal investigations for different organ function (as liver and kidney function).
* Severe pre-eclampsia :40 patients fulfilling anyone or more of the following criteria (The American College of Obstetricians and Gynecologists, 2010)(ACOG):

  * Systolic blood pressure > 160 mmHg
  * Diastolic blood pressure > 110 mmHg (on two occasions at least 6 hours apart while the patient is on bed rest)
  * Proteinuria of 5000mg (5g) or higher on a 24-hour urine collection or at least 3+ on two random urine samples collected at least 4 hours apart
  * Oliguria < 500 mL urine output in 24 hours
  * Cerebral or visual functional disturbances (cns irritability)
  * Pulmonary edema or cyanosis (not due to excessive intravenous volume replacement)
  * Epigastric or right-upper quadrant abdominal pain
  * Impaired liver function on laboratory analysis (elevated aspartate aminotransferase (AST), alanine amino transferase(ALT), or lactate dehydrogenase(LDH))
  * Thrombocytopenia (platelet count < 150,000/uL)
  * Fetal growth restriction.

ELIGIBILITY:
Inclusion criteria:

* pregnant women 3rd trimester
* any age
* medically free at least by history
* signs and or symptoms of pre-eclampsia

Exclusion Criteria:

* Other causes elevate CA-125 as: ovarian cancer, endometrial cancer, breast cancer and benign conditions as: endometriosis and liver cirrhosis.

Chronic hypertension

* Diabetes Mellitus (DM)
* Liver diseases
* Thyroid disorders
* Kidney diseases
* Cardiac diseases

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population comprises pregnant women once diagnosed pre-eclampsia, attending to Ain Shams University Maternity Hospital, or for antinatal care of the corrosponding gestational age.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-07 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
increase serum CA-125 in pre-eclamptic patients | 1 year
  measuring serum CA-125

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Tawfek, Pofessor, Study Director — ain-shams university , cairo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cebesoy FB, Balat O, Dikensoy E, Kalayci H, Ibar Y. CA-125 and CRP are elevated in preeclampsia. Hypertens Pregnancy. 2009 May;28(2):201-11. doi: 10.1080/10641950802601187. PMID 19437230